CLINICAL TRIAL: NCT05812664
Title: The Comparison of Effects of Bolus, Intermittent (Nocturnal Pause) and Continuous Enteral Feeding Methods on Blood Glucose and Feeding Intolerance in ICU Patients With Sepsis, Prospective, Randomized, Controlled Study
Brief Title: The Effects of Bolus, Intermittent and Continuous Enteral Feeding on Blood Glucose and Feeding Intolerance in ICU Patients With Sepsis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Senay Goksu, SPECIALIST, MD, Principal Investigator, Principal Assistant, Umraniye Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: ENTERAL FEEDİNG
Record Dates: First submitted 2023-03-11; First posted 2023-04-14 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Enteral Feeding Intolerance
Keywords: plasma glucose levels,; enteral feeding intolerance; enteral feeding methods; sepsis
MeSH Terms: conditions — Sepsis | interventions — Enteral Nutrition; Blood Glucose

STUDY DESIGN:
Intervention Model Description: If the patients were diagnosed with sepsis in ICU, they were not fed after 24:00, and if the gastric residual measured at 05:00 in the morning was negative, they were included in the study. The patients were examined in 3 groups. The number of samples required to be taken in the power analysis performed (G*power 3.1) was found to be 93 (31 patients in each group) (power value 0.80, alpha error probability=0.05). Patients for the groups were randomly selected by the closed envelope method. A total of 93 envelopes, 31 for each group, were prepared. When the patient was diagnosed with sepsis, if he/she met the inclusion criteria, a random envelope was selected to determine the patient's group. After inclusion in the study, a closed envelope was added again for the patients who should be excluded from the study.
Who Masked: Participant, Outcomes Assessor
Masking Description: Limitation of the study; since the patients were intubated and under sedation, they did not know the diet applied to them, but the physician/nurse who examined the residue and PGD knew the diet. Unfortunately, the person who evaluated these two parameters could not be blinded, as it would not be possible to give without showing the feeding methods. However, groups 1-2-3 were reported to the statistician who analyzed the data. The feeding methods of the groups was not reported.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- bolus feeding group (Experimental): bolus feeding method;The amount of food to be given for 24 hours calculated for the patient was given as 4 equal amounts for 40 minutes at 4 different times. Starting with 150 cc, the target calorie was reached by increasing 100 cc according to the intolerance before the next feeding hour.
  Interventions: Other: enteral feeding; Procedure: blood glucose measurements; Procedure: Evaluation of feeding intolerance with gastric residue
- intermittent feeding group (Experimental): The formula was started as 40 cc/h continuous infusion. It was interrupted after 5 hours. 30 minutes after the break, PGD was measured and intolerance was checked, and if the residue was negative, it was increased by 40 cc. The amount was increased until reaching the amount of formula that should be given for 24 hours calculated for the patient. This cycle was repeated 3 times in 24 hours. At 24:00, it was stopped and feeding was interrupted between 24:00 and 06:00.
  Interventions: Other: enteral feeding; Procedure: blood glucose measurements; Procedure: Evaluation of feeding intolerance with gastric residue
- continous feeding group (Active Comparator): The same method was applied as in Group 2. However, after 24:00, feeding was not interrupted and continued as the 4th cycle.
  Interventions: Other: enteral feeding; Procedure: blood glucose measurements; Procedure: Evaluation of feeding intolerance with gastric residue

INTERVENTIONS:
Other: enteral feeding — The amount of enteral nutrition that should be given daily was calculated by the nutritionist using the Harris-Benedict formula. Formula at room temperature was given with a nasogastric foley catheter and a feeding pump. The position of the nasogastric Foley catheter in the stomach was confirmed by the PAAC graph when it was first inserted, and by listening before each feeding. Feeding was done in a position with the head at 30 degrees.
Procedure: blood glucose measurements — Blood glucose values were measured in all groups at 06:00, 12:00, 18:00 and 24:00, 4 times a day for 7 days. The sample was taken from the patient's cannula and examined in the biochemistry lab. The targeted range in the measurements was accepted as 70-180 mg/dl.
Procedure: Evaluation of feeding intolerance with gastric residue — gastric residue assessment; 30 minutes after the feeding was stopped, the N/G tube was drained and the amount coming 30 minutes later was evaluated. Residue positive was defined as the return of more than half of the amount of formula in the last cycle. The same was continued without increasing the amount given. If the incoming amount was less than half, the residue was evaluated as negative and the formula was continued by increasing the predetermined amount.

SUMMARY:
Comparison of the effects of bolus, intermittent and continuous enteral feeding techniques on plasma glucose level and enteral feeding intolerance in adult intensive care unit patients with sepsis.

DETAILED DESCRIPTION:
in this prospective, controlled trial the main aim is to evaluate the effects of bolus, intermittent and continuous enteral feeding techniques on plasma glucose level in intensive care patients with sepsis diagnosis and to determine whether they are superior to each other in providing norma-glycemia. The secondary aim is to determine the effect of these 3 different enteral feeding techniques on enteral feeding intolerance.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized in ICU for more than 3 days
* Ages between 18-70 years
* APACHI II is in the range of 8-25
* BMI in the range of 18.5-30
* Able to receive enteral nutrition from N/G
* Intubated on ventilator support
* No previous diagnosis of Diabetes Mellitus,
* Those who have not had Gastro intestinal System surgery in the last 6 months
* Patients not receiving inotropic support
* not receiving hemodiafiltration
* No history of allergy to the food used
* Patients with a focus of infection and/or culture-positive patients diagnosed with sepsis according to Q SOFA (cultures were taken from all patients)

Exclusion Criteria:

* patient's death during the study
* Taking more than 40 mg of IV steroids daily
* Increased baseline APACHI II score
* Development of the patient's need for inotropes
* Elimination of inclusion criteria
* negative culture

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
effect of enteral feeding methods on blood glucose levels | for 7 days after the start of feeding
  Evaluation of hypo/hyperglycemia development by measuring blood glucose level 4 times a day

SECONDARY OUTCOMES:
feeding intolerance | during the 7th day with the start of feeding
  effect on feeding intolerance, detection of more than half of the feeding amount will be taken as gastric residue positive so intolerance positive

CONTACTS AND LOCATIONS:
Locations (1):
- Umraniye Education and research hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
all IPD shared with other researches